CLINICAL TRIAL: NCT06623123
Title: Multimodality Smartphone App Delivered Therapy for Tinnitus - a Protocol for a Randomised Controlled Trial
Brief Title: Oto Smartphone App in Treating Tinnitus Amongst Adult Patients Compared with Standard Talking Therapies
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Responsible Party: Principal Investigator, Amir Habeeb, Principal Investigator, East and North Hertfordshire NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RD2023-05 OTO; Corporate Funding (Other: Oto Health Ltd)
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Tinnitus
Keywords: tinnitus; therapeutics; telemedicine; outcomes; otology; otolaryngology
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Masking Description: researchers to data generated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tinnitus Retraining Therapy (TRT) Arm (Active Comparator): Tinnitus-retraining therapy will be offered in the control arm which represents the standard evidence-based intervention on the NHS. (2) Participants enrolled to this arm will undertake tinnitus retraining therapy with a trained audiologist. The sessions will last 30 minutes with the option for further sessions should the patient which to have more support with their tinnitus to mimic the NHS programme as much as possible. These sessions will encompass a brief audiological history followed by therapy tailored to the patient's needs allowing for patient-centred optimisation of tinnitus burden and secondary comorbidities. This may include relaxation, CBT and advice surrounding sound as well as white noise masking therapy.
  Interventions: Behavioral: Tinnitus Retraining Therapy (TRT)
- Oto Smartphone Application (Experimental): The smartphone application delivers personalized tinnitus therapy combining evidence-based CBT with mindfulness, patient education as well as physical therapy such as stretches and exercises. There are additional sounds available to listen to from the sound library. There will be a structured programme that the participants can work through however they are encouraged to personalise their own therapy.
  Interventions: Device: Oto Smartphone Application (Oto Health Ltd)

INTERVENTIONS:
Device: Oto Smartphone Application (Oto Health Ltd) — The smartphone application delivers personalized tinnitus therapy combining evidence-based CBT with mindfulness, patient education as well as physical therapy such as stretches and exercises. There are additional sounds available to listen to from the sound library. There will be a structured programme that the participants can work through however they are encouraged to personalise their own therapy.
  Arms: Oto Smartphone Application
Behavioral: Tinnitus Retraining Therapy (TRT) — Tinnitus-retraining therapy will be offered in the control arm which represents the standard evidence-based intervention on the NHS. (2) Participants enrolled to this arm will undertake tinnitus retraining therapy with a trained audiologist. The sessions will last 30 minutes with the option for further sessions should the patient which to have more support with their tinnitus to mimic the NHS programme as much as possible. These sessions will encompass a brief audiological history followed by therapy tailored to the patient's needs allowing for patient-centred optimisation of tinnitus burden and secondary comorbidities. This may include relaxation, CBT and advice surrounding sound as well as white noise masking therapy.
  Arms: Tinnitus Retraining Therapy (TRT) Arm

SUMMARY:
A study that looks at treating tinnitus and its associated burden, insomnia and quality of life effects with a smartphone app when compared with the talking therapies already offered on the national health service. Three separate questionnaires will be used to collect this data from patients at regular time intervals.

DETAILED DESCRIPTION:
Single-site randomised controlled study looking at tinnitus burden, insomnia severity and quality of life in adults with chronic primary subjective tinnitus when using Oto smartphone app compared with National Institute for Health and Care Excellence (NICE) approved tinnitus retraining therapy. This will be assessed objectively through questionnaires at the baseline meeting, one month, three months and six months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (male or female) aged over 18 years of age presenting to NHS ENT and hearing services with primary non-pulsatile tinnitus irrespective of hearing.
* Patients must be suffering from tinnitus for a minimum of 3 months
* Patients that have a willingness to use as well as have access to a smartphone device capable of running Oto.
* Willing and able to provide written informed consent.
* Those that would be offered tinnitus retraining therapy (TRT) as management for their primary tinnitus

Exclusion Criteria:

* Patients with secondary tinnitus as confirmed by magnetic resonance imaging (MRI).
* Patients undergoing any other tinnitus therapies concurrently (including hearing aids / implants). Previous tinnitus therapies including CBT in the past are accepted.
* Patients who are not willing to use the app due to not having a suitable phone to download the application or due to own limitations in working Oto.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Burden | 6 months total post intervention start date
  Tinnitus burden via Tinnitus Functional Index questionnaires at 0 months (T0), 1 month (T1), 3 months (T2) and 6 months (T3).

SECONDARY OUTCOMES:
Insomnia Severity | 6 months total post intervention start date
  Insomnia index as calculated via Insomnia Severity Index questionnaire at 0 months (T0), 1 month (T1), 3 months (T2) and 6 months (T3).
Quality of Life | 6 months total post intervention start date
  Quality of life as calculated via the WHO Quality of Life - BREF questionnaire at 0 months (T0), 1 month (T1), 3 months (T2) and 6 months (T3).

CONTACTS AND LOCATIONS:
Locations (1):
- East and North Hertfordshire NHS Trust, Stevenage, Hertfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Vahedi S. World Health Organization Quality-of-Life Scale (WHOQOL-BREF): Analyses of Their Item Response Theory Properties Based on the Graded Responses Model. Iran J Psychiatry. 2010 Fall;5(4):140-53. PMID 22952508
- [Background] Carlbring P, Andersson G, Cuijpers P, Riper H, Hedman-Lagerlof E. Internet-based vs. face-to-face cognitive behavior therapy for psychiatric and somatic disorders: an updated systematic review and meta-analysis. Cogn Behav Ther. 2018 Jan;47(1):1-18. doi: 10.1080/16506073.2017.1401115. Epub 2017 Dec 7. PMID 29215315
- [Background] Mehdi M, Dode A, Pryss R, Schlee W, Reichert M, Hauck FJ. Contemporary Review of Smartphone Apps for Tinnitus Management and Treatment. Brain Sci. 2020 Nov 17;10(11):867. doi: 10.3390/brainsci10110867. PMID 33212928
- [Background] Lewis S, Chowdhury E, Stockdale D, Kennedy V; Guideline Committee. Assessment and management of tinnitus: summary of NICE guidance. BMJ. 2020 Mar 31;368:m976. doi: 10.1136/bmj.m976. No abstract available. PMID 32234748
- [Background] Shargorodsky J, Curhan GC, Farwell WR. Prevalence and characteristics of tinnitus among US adults. Am J Med. 2010 Aug;123(8):711-8. doi: 10.1016/j.amjmed.2010.02.015. PMID 20670725
- See also: Randomiser — https://www.sealedenvelope.com/randomisation